CLINICAL TRIAL: NCT05898412
Title: Retrospective Real World Evidence Study to Describe Characteristics and Outcomes in Dutch Patients Admitted to the Hospital With a Factor Xa Inhibitor-associated Bleeding Treated With Andexanet Alfa
Brief Title: Retrospective Study on Characteristics and Outcomes in Hospitalised Patients Treated With Ondexxya
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: LOGEX Healthcare Analytics Amsterdam The Netherlands (Unknown)
Responsible Party: Sponsor
Other Study IDs: D9603R00007
Record Dates: First submitted 2023-04-06; First posted 2023-06-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhage
Keywords: Observational; Retrospective; Major bleeding; Andexanet alfa; Factor Xa inhibitor; Patient characteristics; Treatment strategy; Outcomes
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Andexanet alfa: Hospitalized patients treated with andexanet alfa
  Interventions: Drug: Andexanet alfa
- Thrombotic Event: Hospitalized patients treated with andexanet alfa who experienced a thrombotic event (TE) within 30 days
  Interventions: Drug: Andexanet alfa

INTERVENTIONS:
Drug: Andexanet alfa — Patients treated with andexanet alfa

SUMMARY:
This is an observational retrospective database study of hospitalized patients treated with andexanet alfa in approximately 10 Dutch hospitals. Currently there is limited information on the patient characteristics and outcomes of patients who are treated with andexanet alfa in The Netherlands and how it is used. This is of interest for treating clinicians because there is a need for a patient profile, also due to the on par position of andexanet alfa with PCC in the Dutch national guideline.

Analysis of the data showed that 14 patients of the 218 patients included in the study (6.4%) experienced a thrombotic event (TE) within 30 days after treatment with andexanet alfa. The protocol was amended to allow for an in depth analysis of the 14 TE cases.

DETAILED DESCRIPTION:
The direct oral anticoagulants (DOAC) rivaroxaban and apixaban inhibit factor Xa (FXa) and are widely used in clinical practice, due to the ease of administration, lack of need for frequent monitoring and dose adjustment and an improved safety profile. However, reversal of the anticoagulant effect of these FXa inhibitors (FXai) can be acutely required in case of serious bleeding events, like intracranial hemorrhage (ICH).

Ondexxya® (andexanet alfa) has been approved and is available in the Netherlands since 2019. Andexanet alfa is a modified FXa with no coagulant activity. It has a high binding affinity to DOACs and can therefore be used as reversal agent against DOACs. However, andexanet alfa is not used in all Dutch centers. In some hospitals, instead of andexanet alfa, nonspecific agents are used to manage FXai-associated ICH bleeding, like four-factor prothrombin complex concentrate (4F-PCC).

Due to the on par position of andexanet alfa and 4F-PCC in the Dutch multidisciplinary antithrombotic guideline, there is no clear patient profiling for the use of andexanet alfa for Dutch clinicians.

The lack of randomized clinical trials comparing the efficacy and safety of andexanet alfa and 4F-PCC also does not help to provide clarity. There is real world evidence data available (Coleman et al. 2020; Cohen et al. 2022; Costa et al. 2022) but these studies uses data from the US and the UK, and consistently report a superior effectiveness of andexanet alfa over 4F-PCC. However, there is considerable variation in the reported effectiveness between these studies, with mortality rate ranging from 4% to 15.3%. Potentially, differences in methodology and sample size, in addition to patient populations and bleeding locations varying between analyses, have resulted in this variation. Additionally, anecdotal information indicates that in some cases andexanet alfa is administered after 4F-PCC fails.

Therefore, the aim of the present analysis is to characterize the patient population that received andexanet alfa in the Dutch healthcare system. Also, we aim to describe clinical outcomes in patients treated with andexanet alfa in daily clinical practice in the Netherlands.

Providing real world data on the patient characteristics and outcomes of andexanet alfa treated patients in the Netherlands, may support clinicians in the future identification of the patient who benefit most of treatment with andexanet alfa.

The protocol was amended to allow for an in-depth analysis of the 14 individual cases who experienced a TE within 30 days after treatment with andexanet alfa, in order to establish the temporal relationships and clinical impact/outcome of this event on the patient, stratified by risk factors for the occurrence and outcome of the TE.

The results will be shown in a 'swimmers plot', showing the events relative to the onset of the major bleed and the clinical outcome of the TE, including risk classification based on the presence of co-morbidities and several risk factors such as TE and HF in medical history, weight/BMI, BP, restart DOAC, info on initial hemostasis, ICH/Chadvasc score, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Received at least one dose of andexanet alfa

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients >18 years of age treated with at least one dose of andexanet alfa
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Patient characteristics | Baseline (which is the date andexanet alfa is administered, i.e. indexdate)
  At baseline the following patient characteristics will be described: age, sex, type of bleeding (ICH, GI or other), concomittant medication, FXai indication, type and dose, comorbidities, GCS at admission (for ICH only), eGFR and Hb, type of hospital.
  For 14 TE cases: weight, BMI anti-FXa level, type of blood transfusion, baseline haematoma volume (ICH only), bloodpressure parameters (initial, 1 hr, 2 hr, mean arterial pressure, 24hr control), pulse, noradrenalin, ICH score/Chadvasc score, do not resuscitate status, info on initial hemostasis that could inform on prognosis (if available from CT) will be described

SECONDARY OUTCOMES:
Andexanet alfa dose | Baseline
  Dose of andexanet alfa in mg
Time from symptom onset to hospital admission | Baseline
  time between the onset of the bleeding symptoms to admission to the hospital in hours
Time from symptom onset to andexanet alfa administration | Baseline
  Time between onset of bleeding symptoms to start of the treatment with andexanet alfa in hours
Time between last dose of FXai and andexanet alfa administration | Baseline
  Time between last dose of FXai taken by the patient and the start of the treatment with andexanet alfa in hours
Frequency that andexanet alfa is administered before or after replacement therapy; | Baseline
  Number of times that a patient is treated with andexanet alfa in combination with replacement therapy
Time interval between replacement therapy and andexanet alfa administration | Baseline
  Time between treatment with andexanet alfa and replacement therapy in hours

OTHER OUTCOMES:
Cumulative incidence of thrombotic events | from index date to maximum 30 days FU
  Thrombotic events leading to (re-)hospitalization within 30 days after andexanet alfa treatment; thrombotic events occurring during the hospitalization for the index bleeding
  For 14 TE cases, the basis of the TE diagnosis (e.g. procedure, radiology, clinic, symptoms, lab etc) and the impact/outcome parameter of the TE will be described based on available information in the free text in EPD, varying from 'no impact' and 'severe impact' to 'death'
Inpatient mortality | from index date to maximum 30 days FU
  Inpatient mortality within 30 days after andexanet alfa treatment
  For 14 TE cases, the cause of death and wether it was caused by a decision to terminate treatment will be described
Rehospitalization | from index date to maximum 30 days FU
  All rehospitalizations (including diagnosis) within 30 days after andexanet alfa treatment
Length Of Stay (LOS) | from index date to maximum 30 days FU
  Total LOS and ICU LOS in days.
  These will be aggregated with the number of (i) surgical interventions to treat the bleeding,(ii) mechanical ventilation/intubation, (iii) brain CTs and MRIs and (iv) endoscopies to estimate the health care resource use
Number of surgical interventions | from index date to maximum 30 days FU
  Number of times that a surgical intervention is needed to treat the bleeding
  These will be aggregated with (i) LOS/ICU LOS and the the number of (ii) mechanical ventilation/intubation, (iii) brain CTs and MRIs and (iv) endoscopies to estimate the health care resource use
Number of mechanical ventilation/intubation | from index date to maximum 30 days FU
  Number of times that a patient is intubated/ventilated mechanically
  These will be aggregated with (i) LOS/ICU LOS and the the number of (ii) surgical interventions (iii) brain CTs and MRIs and (iv) endoscopies to estimate the health care resource use
Number of CT scans and MRI's | from index date to maximum 30 days FU
  Number of CT scans and MRIs needed to diagnose the bleeding
  These will be aggregated with (i) LOS/ICU LOS and the the number of (ii) surgical interventions (iii) mechanical ventilation/intubation and (iv) endoscopies to estimate the health care resource use
Number of endoscopies | from index date to maximum 30 days FU
  Number of times that a an endoscopy is performed to diagnose/treat bleeding
  These will be aggregated with (i) LOS/ICU LOS and the the number of (ii) surgical interventions (iii) mechanical ventilation/intubation and (iv) brain CTs and MRIs to estimate the health care resource use
Type of anti-coagulant re-initiated after indexdate | from index date to maximum 30 days FU
  Type of any anti-coagulant that is reinitiated after index date
Timing of any anti-coagulant re-initiated after index date | from index date to maximum 30 days FU
  Timing of any anti-coagulant that is reinitiated after index date in days
Dose of any anti-coagulant re-initiated after index date | from index date to maximum 30 days FU
  Dose of any anti-coagulant that is reinitiated after index date in mg
anticoagulant indication and dose, surgery activity date, andexanet alfa administration date | baseline
  To describe if andexanet alfa is administered to patients treated with edoxaban, enoxaparin or other anticoagulant or prior to acute surgery as primary indication
Anti factor Xa activity measurement activities and results and timing of andexanet alfa adminstration | Baseline
  To describe if measurement of anti factor Xa activity prior to andexanet alfa administration is performed, and if results are available in time to impact clinical decision making
Doselevel of andexanet alfa | Baseline
  it will be described whether the doselevel of andexanet alfa in mg, is related to the time between the last FXai administration and hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman CI, Dobesh PP, Danese S, Ulloa J, Lovelace B. Real-world management of oral factor Xa inhibitor-related bleeds with reversal or replacement agents including andexanet alfa and four-factor prothrombin complex concentrate: a multicenter study. Future Cardiol. 2021 Jan;17(1):127-135. doi: 10.2217/fca-2020-0073. Epub 2020 Jul 3. PMID 32618210
- [Background] Costa OS, Connolly SJ, Sharma M, Beyer-Westendorf J, Christoph MJ, Lovelace B, Coleman CI. Andexanet alfa versus four-factor prothrombin complex concentrate for the reversal of apixaban- or rivaroxaban-associated intracranial hemorrhage: a propensity score-overlap weighted analysis. Crit Care. 2022 Jun 16;26(1):180. doi: 10.1186/s13054-022-04043-8. PMID 35710578
- [Background] Cohen AT, Lewis M, Connor A, Connolly SJ, Yue P, Curnutte J, Alikhan R, MacCallum P, Tan J, Green L. Thirty-day mortality with andexanet alfa compared with prothrombin complex concentrate therapy for life-threatening direct oral anticoagulant-related bleeding. J Am Coll Emerg Physicians Open. 2022 Mar 5;3(2):e12655. doi: 10.1002/emp2.12655. eCollection 2022 Apr. PMID 35280921